CLINICAL TRIAL: NCT00994604
Title: The Effects of Broccoli Sprout Extract on Obstructive Lung Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Robert Brown, Professor, Johns Hopkins University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RB-001
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Results first posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2016-12

CONDITIONS: Asthma; COPD
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- broccoli sprout extract (Experimental): This a before and after treatment study. The subjects will consumer broccoli sprout extract (BSE) for two weeks (14d). Lung function and Chest CT will be performed before and after BSE consumption.
  Interventions: Drug: broccoli sprout extract

INTERVENTIONS:
Drug: broccoli sprout extract — consumption of broccoli sprout extract for 2 weeks

SUMMARY:
The purpose of this study is to examine whether broccoli sprout extract can effect lung function measurements in individuals with asthma and COPD.

DETAILED DESCRIPTION:
Asthma afflicts 23 million people, results in nearly 13 million ambulatory physician encounters, and 440,000 hospitalizations annually. The economic burden for 2010 is estimated to run $20.7 billion.

Although steroids are the mainstay of treatment, they do not "cure" the disease. While inflammation may be the inciting factor, other mechanisms must play a crucial role in this process. Elevated oxidative stress could cause the kind of chronic inflammation associated with asthma, and could provide an explanation for recurrent asthma attacks. Cigarette smoke, both primary and secondary exposure, worsens the oxidative stress balance in the airways. Thus, the continuing focus on simply treating the inflammation is a barrier to progress. It is critical to examine other factors, such as abnormal oxidative stress through specific pathways that may affect airway inflammation and asthma attacks.

One compound, that repairs oxidative stress pathways, is sulforaphane, a food compound found in vegetables, including broccoli sprouts. Preliminary data demonstrate that broccoli sprout extract (BSE), rich in sulforaphane, improves airflow measures in asthmatics.

We plan to examine whether the airflow abnormalities in asthma, and the exacerbation from cigarette smoke, can be prevented by the administration of BSE, and determine the primary inflammatory and oxidative stress signaling pathways involved in the protection provided by BSE.

ELIGIBILITY:
Inclusion Criteria:

* asthma
* COPD

Exclusion Criteria:

* currently on chronic oral steroid medications
* current respiratory symptoms
* pregnant
* FEV1 less than 40% predicted at baseline
* extreme degrees of bronchial hyperreactivity
* recent respiratory infection (<3 weeks)
* unstable symptoms in the prior month
* a history of intubation for respiratory symptoms within the past year
* any history of cardiac disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Brown, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Medical Institutions, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
This was a pilot study.

RESULTS

PARTICIPANT FLOW:
Groups:
- Broccoli Sprout Extract: pre- and post-consumption of broccoli sprout extract for 2 weeks
Period: Overall Study
Arm/Group | Broccoli Sprout Extract
Started | 51
Completed | 45
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Broccoli Sprout Extract
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (13)
Gender [Count of Participants; unit: Participants]
  Female | 29
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome is the Change in Bronchodilation and Bronchoprotection After Broccoli Sprout Extract
Description: Bronchodilator index = (1- ((1 - ((forced expiratory volume in 1 second after Methacholine A and after Deep Inspiration )÷( forced expiratory volume in 1 second baseline)))÷ (1 - ((forced expiratory volume in 1 second after Methacholine)÷( forced expiratory volume in 1 second baseline)))))x100
  Bronchoprotection index = (1- ((1 - ((forced expiratory volume in 1 second after Deep Inspirations and after Methacholine B )÷( forced expiratory volume in 1 second baseline B)))÷(1 - ((forced expiratory volume in 1 second after Methacholine A)÷( forced expiratory volume in 1 second baseline A))))) x 100
Time Frame: baseline and two weeks
Measure: Mean (Standard Deviation); unit: index
Groups:
- Broccoli Sprout Extract - BP; Broccoli Sprout Extract - BD: pre- and post-consumption of broccoli sprout extract for 2 weeks
Arm/Group | Broccoli Sprout Extract - BP | Broccoli Sprout Extract - BD
Number analyzed (Participants) | 45 | 45
index | 10.3 (57.1) | 26.7 (30.6)

2. Secondary Outcome: Changes in Airway Size by Computed Tomography
Description: Changes in size airways as measured by computed tomography
Time Frame: baseline and after two weeks
Measure: Mean (Standard Deviation); unit: size in mm^2
Groups:
- Airway Size Pre BSE; Airway Size Post BSE: CT scan measurements of changes in luminal area with BSE treatment measured at either total lung capacity (TLC) or functional residual capacity (FRC) (mean ± SD).
Arm/Group | Airway Size Pre BSE | Airway Size Post BSE
Number analyzed (Participants) | 45 | 45
size in mm^2 | 30.9 (1.8) | 32 (4.5)

ADVERSE EVENTS:
Time Frame: entire study
Arm/Group | Broccoli Sprout Extract
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No